CLINICAL TRIAL: NCT05829317
Title: Parenteral Magnesium Prophylaxis for the Prevention of New-Onset Atrial Fibrillation in Critically Ill Patients - a Pilot Feasibility Study
Brief Title: Magnesium Prophylaxis for the Prevention of New-Onset Atrial Fibrillation in Critically Ill Patients
Acronym: ATOMIC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Stephanie Sibley (Other)
Collaborators: Southeastern Ontario Academic Medical Organization (SEAMO) (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Stephanie Sibley, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ATOMIC
Record Dates: First submitted 2023-03-15; First posted 2023-04-25 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness; New Onset Atrial Fibrillation
Keywords: Prophylaxis; Prevention
MeSH Terms: conditions — Critical Illness | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium Sulfate (Experimental): 4g Magnesium sulfate (100mL) BID, given intravenously over 2 hours, for a total of 10 doses
  Interventions: Drug: Magnesium sulfate
- 0.9% NaCl (Placebo Comparator): 100mL 0.9% NaCl BID, given intravenously over 2 hours, for a total of 10 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium sulfate — Intravenous Magnesium sulfate
  Arms: Magnesium Sulfate
Drug: Placebo — 0.9% NaCl
  Arms: 0.9% NaCl

SUMMARY:
A double-blind, multi-centre, randomized, placebo-controlled, feasibility pilot trial in the prevention of new onset atrial fibrillation of critically ill patients admitted to an ICU.

DETAILED DESCRIPTION:
Most studies of new onset atrial fibrillation (NOAF) in critical illness focus on treatment of this arrhythmia but this innovative study will focus on prevention. Parenteral Mg is a low cost and readily available treatment that may be beneficial for reducing the incidence of NOAF in critically ill patients, with the potential to improve patient centred outcomes and provide a cost effective prophylaxis. The main outcome of this study is to determine if it is feasible to conduct a randomized controlled trial comparing parenteral magnesium sulfate with placebo for the prophylaxis of new onset atrial fibrillation in critically ill patients.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years;
2. Admitted to an ICU with one or more of the following:

   1. Non-invasive ventilation (including CPAP, Bipap and high flow oxygen (>10L/min) or invasive mechanical ventilation with an expected duration >24 hours for respiratory failure (hypercarbic or hypoxic)
   2. Vasopressor or inotropic support with an expected duration of >24 hours
   3. Cardiac arrest
3. Continuous cardiac monitoring.

Exclusion Criteria

1. Receiving ICU intervention (Non-invasive ventilation (including high flow nasal canula), invasive mechanical ventilation or inotropic support) for >18 hours
2. Receiving IMV for airway protection only (for example, isolated head trauma)
3. Active atrial fibrillation at the time of enrolment
4. On oral or continuous infusion of Amiodarone
5. Unlikely to survive >24 hours or palliative patients
6. Cardiac surgery patients
7. Patients requiring parenteral magnesium therapy (e.g. pre-eclampsia, asthma)
8. Patients receiving dialysis
9. Positive pregnancy test (females <50 years old)
10. Previously enrolled in this trial
11. Treating physician refuses enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
RCT Feasibility | 90 days
  To assess feasibility of patient recruitment, randomization procedures, intervention and data collection and measure protocol adherence. Protocol adherence ≥ 90% (We define protocol adherence as administration of first dose of study drug within 18 hours (+1hr window) of 1st ICU intervention (life sustaining therapy) delivery of all additional
RCT Feasibility | 90 days
  Recruitment rate of ≥ 2 patients/month/ICU

SECONDARY OUTCOMES:
Equipoise and Feasibility | 365 days
  Physician willingness to recruit patients in the setting of existing electrolyte replacement protocols; effectiveness of blinding; proportion of patients who meet eligibility criteria of those admitted to ICU; proportion of eligible patients for whom consent is obtained; proportion of patients who re-consent when they regain capacity for those randomized under the deferred consent model; proportion of patients lost to follow-up; time for research personnel to complete study related tasks.
Acute Care Outcomes | 28 days
  Total number of patients developing AF within 28 days of enrolment (AF will be defined as at least 30 seconds of NOAF detected by cardiac monitoring or ECG); Use of rate and rhythm controlling agents, vasoactive agents, diuretics, steroids, anticoagulants, bleeding events, thromboembolic events (as defined in the 2018 Canadian Stroke Best Practices Guideline1; these will be adjudicated by a neurologist blinded to study groups), persistent organ dysfunction, mortality
Hospital Outcomes | 28 days
  Days alive and ventilator free, ICU length of stay, and hospital length of stay.
Adverse Events | 28 days
  Adverse drug reactions including bradycardia (HR <60 bpm); severe bradycardia (HR <50 bpm); clinically significant bradycardia (bradycardia requiring inotropes, vasopressors, external pacing, temporary pacemaker, or discontinuation of the trial medication); hypotension (MAP< 65mmHg, or systolic blood pressure [SBP]>20mmHg below admission baseline); clinically significant hypotension (hypotension requiring vasopressors, fluid administration, or discontinuation of the trial medication) while the study drug is being infused.
Functional Outcomes | 365 days
  EQ-5D score, death after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sibley, MD, Principal Investigator — Queen's University
Locations (4):
- Canada (4):
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Undecided